CLINICAL TRIAL: NCT05195125
Title: Phase I Clinical Trial Utilizing Direct Peritoneal Resuscitation in Liver Transplant Recipient Population at Increased Risk of Return to the Operating Room and Early Allograft Dysfunction
Brief Title: Use of Direct Peritoneal Resuscitation in High-risk Liver Transplant Recipients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-4214
Record Dates: First submitted 2021-12-14; First posted 2022-01-18 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: End Stage Liver DIsease; Obesity; Acute Kidney Injury
Keywords: Liver transplant; Obesity; Renal failure
MeSH Terms: conditions — End Stage Liver Disease; Obesity; Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: All study subjects will be enrolled to the treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Direct Peritoneal Resuscitation (DPR) Group (Experimental): At the time of abdominal closure and determination that the patient will either go to extended stay or the intensive care unit, three drains will be placed per standard of care. An additional 19 French drain will be placed at the ligament of Treitz at the base of the mesentery. Following abdominal closure DPR will be initiated with commercially available 2.5% glucose-based peritoneal dialysis solution at a rate of 1.5 cc/kg/hr based on previously reported therapy in trauma. Drains will be connected to continuous wall suction. This infusion will continue for the duration the patients stay in extended stay (8 hours) if they are deemed eligible for hospital ward admission, or for 24 hours if requiring ICU care. These patients will then be observed for their hospital course and monitored for outcomes listed above.
  Interventions: Procedure: Direct Peritoneal Resuscitation

INTERVENTIONS:
Procedure: Direct Peritoneal Resuscitation — Direct peritoneal resuscitation involves the abdominal infusion and drainage of a peritoneal dialysate in high-risk liver transplant patients, for up to 24 hours after surgery.

SUMMARY:
This study is being conducted to assess the safety of Direct Peritoneal Resuscitation (DPR) in high-risk liver transplant patients. The investigators want to also identify if this method of recovery after large surgery has the same benefits in liver transplant patients as have been appreciated in other surgical patients. The combination of elevated BMI and impaired kidney function increases the risk of 1) needing intensive care unit (ICU) admission after surgery, 2) slow function of the new liver [technically termed Early Allograft Dysfunction (EAD)] and 3) need for more than one operation. The study team also aims to identify if DPR can reduce these risks and not cause other unexpected complications following surgery. DPR involves the infusion of a solution into the abdomen and has been shown to reduce edema and improve blood flow in organs. The solution used in this study is a commercially available peritoneal dialysate, a dextrose containing solution that is infused into the abdominal cavity and is routinely used in patients with end-stage renal disease requiring dialysis.

DETAILED DESCRIPTION:
The central hypothesis of this study is that direct peritoneal resuscitation is a safe therapy following liver transplantation and is associated with a reduced rate of return to the operating room.

AIM 1: Determine the safety profile of direct peritoneal resuscitation on liver transplant recipients at risk of return to the operating room and ICU admission. Hypothesis: Liver transplant recipients that receive DPR will have comparable complication rates to historic controls of liver transplant recipients with similar demographics.

AIM 2: Identify if direct peritoneal resuscitation demonstrates a trend towards a reduced rate of return to the operating room compared to historic controls. Hypothesis: DPR will demonstrate a trend of a reduce rate of return to the operating room of liver transplant patients after index operation compared to historic controls.

AIM 3: Identify if direct peritoneal resuscitation reduces the rate of early allograft dysfunction and other organ failure following liver transplantation with interval improvement in post-operative fibrinolysis activity. Hypothesis: DPR will reduce the rate of EAD of liver transplant patients compared to historic controls and is associated with increased fibrinolysis in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Adult liver transplant recipients ≥18 y/o
* Ability to consent
* Pre-operative Creatinine ≥1.1 (or on dialysis) and BMI ≥30

Exclusion Criteria:

* Diaphragmatic injury
* Active spontaneous bacterial peritonitis (SBP) with initiation of antibiotic treatment within 72 hours of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percent of patients that complete DPR infusion without reaching stopping criteria | Up to 24 hours after initiation of direct peritoneal resuscitation

SECONDARY OUTCOMES:
Rate of return to the operating room after index operation | Up to 7 days after transplant
  Amount of patients that require a re-operation after their transplant
Abdominal compartment syndrome requiring reoperation | Events that occur during the duration of the DPR infusion, which will last no more than 24 hours after the participant's transplant surgery.
  Number of patients that develop increased intraabdominal pressure as a consequence of dialysate infusion
Percent of patients that complete DPR infusion | Up to 24 hours after initiation of DPR
Percent of patients that are transferred to hospital ward | Up to 24 hours after surgery
  Patients that are admitted to the hospital ward after surgery, not requiring ICU admission
Rate of early allograft dysfunction | Up to 7 days after transplant
  Patients who experience slow function of their transplanted liver after their transplant
Number of blood product units required during first 24 hours postoperatively | Up to 24 hours after transplant
  The study team will record the number of units of blood product (i.e. "bags" of red blood cells, platelets, etc.) required by the participant in the first day after liver transplantation.
Number of participants that require renal replacement therapy (i.e. hemodialysis) during the first 7 days after liver transplant. | Up to 7 days after transplant
  Researches will record whether the participant developed renal failure requiring renal replacement therapy (i.e. hemodialysis)
Hourly urine output for first 24 hours | Up to 24 hours after transplant
Rate of early infection after transplant | <7 days postoperatively
  Researchers will record any infections that participants develop after transplantation. These may include abscess, peritonitis, bacteremia, and pneumonia.
Rate of late infection after transplant | 7-30 days postoperatively
  Researchers will record any infections that participants develop after transplantation. These may include abscess, peritonitis, bacteremia, and pneumonia.
Rate of mechanical bowel obstruction | Up to 30 days after transplant
  Constipation caused by compression from inside or outside of the bowel lumen
Ileus/time to oral intake | Up to 30 days after transplant
  Time to return of normal bowel function and food tolerance after transplant
Duration of insulin infusion post-operatively | Up to 7 days after transplant
  Insulin requirements after transplant surgery
Ventilator free days | Up to 28 days post-op
  Outcome measurement that looks into rate of respiratory failure requiring prolonged mechanical ventilation after transplant surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hunter B Moore, M.D., P.hD., Principal Investigator — University of Colorado School of Medicine
Locations (1):
- UCHealth - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weaver JL, Smith JW. Direct Peritoneal Resuscitation: A review. Int J Surg. 2016 Sep;33(Pt B):237-241. doi: 10.1016/j.ijsu.2015.09.037. Epub 2015 Sep 16. PMID 26384838
- [Background] Smith JW, Garrison RN, Matheson PJ, Franklin GA, Harbrecht BG, Richardson JD. Direct peritoneal resuscitation accelerates primary abdominal wall closure after damage control surgery. J Am Coll Surg. 2010 May;210(5):658-64, 664-7. doi: 10.1016/j.jamcollsurg.2010.01.014. PMID 20421025
- [Background] Zakaria el R, Garrison RN, Kawabe T, Harris PD. Direct peritoneal resuscitation from hemorrhagic shock: effect of time delay in therapy initiation. J Trauma. 2005 Mar;58(3):499-506; discussion 506-8. doi: 10.1097/01.ta.0000152892.24841.54. PMID 15761343
- [Background] Smith JW, Ghazi CA, Cain BC, Hurt RT, Garrison RN, Matheson PJ. Direct peritoneal resuscitation improves inflammation, liver blood flow, and pulmonary edema in a rat model of acute brain death. J Am Coll Surg. 2014 Jul;219(1):79-87. doi: 10.1016/j.jamcollsurg.2014.03.045. Epub 2014 Apr 5. PMID 24952444
- [Background] Weaver JL, Matheson PJ, Hurt RT, Downard CD, McClain CJ, Garrison RN, Smith JW. Direct Peritoneal Resuscitation Alters Hepatic miRNA Expression after Hemorrhagic Shock. J Am Coll Surg. 2016 Jul;223(1):68-75. doi: 10.1016/j.jamcollsurg.2016.03.024. Epub 2016 Mar 26. PMID 27345902
- [Background] Smith JW, Matheson PJ, Morgan G, Matheson A, Downard C, Franklin GA, Garrison RN. Addition of direct peritoneal lavage to human cadaver organ donor resuscitation improves organ procurement. J Am Coll Surg. 2015 Apr;220(4):539-47. doi: 10.1016/j.jamcollsurg.2014.12.056. Epub 2015 Feb 9. PMID 25797737
- See also: Direct Peritoneal Resuscitation: A review. — https://pubmed.ncbi.nlm.nih.gov/26384838/
- See also: Direct peritoneal resuscitation accelerates primary abdominal wall closure after damage control surgery. — https://pubmed.ncbi.nlm.nih.gov/20421025/
- See also: Direct peritoneal resuscitation from hemorrhagic shock: effect of time delay in therapy initiation. — https://pubmed.ncbi.nlm.nih.gov/15761343/
- See also: Direct peritoneal resuscitation improves inflammation, liver blood flow, and pulmonary edema in a rat model of acute brain death. — https://pubmed.ncbi.nlm.nih.gov/24952444/
- See also: Direct Peritoneal Resuscitation Alters Hepatic miRNA Expression after Hemorrhagic Shock. — https://pubmed.ncbi.nlm.nih.gov/27345902/
- See also: Addition of direct peritoneal lavage to human cadaver organ donor resuscitation improves organ procurement. — https://pubmed.ncbi.nlm.nih.gov/25797737/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05195125/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT05195125/ICF_001.pdf